CLINICAL TRIAL: NCT00413764
Title: A Multicenter, Randomized, Double-Blind, Double Dummy Trial to Compare the Effects Tibolone and Transdermal Continuous Combined Estradiol/Norethisterone on Sexual Desire and Arousal in Postmenopausal Women With Sexual Dysfunction
Brief Title: Efficacy of Tibolone Versus Transdermal E2/NETA on Sexual Function in Naturally Postmenopausal Women (P06089)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06089; C-1774
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — tibolone; estradiol, norethisterone, testosterone drug combination; estradiol, norethindrone drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): tibolone
  Interventions: Drug: tibolone
- 2 (Active Comparator): transdermal continuous combined E2-NETA (estradiol-norethisterone)
  Interventions: Drug: estradiol-norethisterone

INTERVENTIONS:
Drug: tibolone — tibolone (2.5 mg) over 24 weeks
  Other Names: Livial®
  Arms: 1
Drug: estradiol-norethisterone — transdermal continuous combined E2-NETA (estradiol-norethisterone 50/140 mcg) over 24 weeks
  Other Names: Combipatch®; Estalis®
  Arms: 2

SUMMARY:
Tibolone has been registered for treatment of menopausal symptoms. It is, however, not known what the effects are of tibolone in postmenopausal women diagnosed with sexual dysfunction. This is important because there is currently no approved treatment of libido problems in postmenopausal women. Therefore, the primary aim of this study was to compare the effects of tibolone with an estrogen/progestogen skin patch in postmenopausal women diagnosed sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy postmenopausal women, >=48 and <=68 years of age, with an intact uterus.
* Women were to suffer from decreased satisfactory sexual activity compared to younger age and sexual problems were not to be considered caused by relationship/partner problems. The decreased sexual functioning was to result in sexually related personal distress as confirmed by the FSDS (score =15).
* An affirmative answer was to be given to the following questions: (a) In previous years did you find sexual activity satisfying? (b) Has there been a decline in your satisfaction with sexual activity? (c) Are you satisfied with your partner as a friend?
* All subjects were to have an established sexual relationship of at least 6 months duration prior to screening.
* Women were to be sexually active.
* Normal mammography within 6 months prior to randomization.
* Body mass index >18 and <=32 kg/m2.
* Voluntary written informed consent

Exclusion Criteria:

* Any unexplained abnormal uterine bleeding
* Double layer endometrial thickness >4 mm
* Tibolone or transdermal E2/NETA use within 3 months prior to screening
* Progestogen implants or injections and estrogen/progestogen injectable therapy within 6 months prior to screening
* Use of intra-uterine progestogen
* Unsuccessful previous treatment with androgens or compounds known to enhance androgenic activity
* Current successful treatment with androgens, without applying the applicable washout period of 3 months prior to screening
* Any previous or current unopposed estrogen administration, prior use of estrogen pellets or tamoxifen citrate (previous low dose vaginal estrogen-only applications are allowed)
* Use of anti -androgens within the preceding 5 years prior to screening.
* Women with significant organic disorder of sexual dysfunction or a partner with sexual dysfunction
* Women who had early onset sexual dysfunction (>15 years prior to menopause)
* Women suffering from androgenic alopecia, acne or hirsutism
* Women suffering from illnesses influencing sexuality
* Women using medication influencing sexuality
* Moderate to severe depression
* Current or prior use of antidepressant within 8 weeks prior to screening
* Major gynecological surgery in the preceding 3 months
* Any serious disease or disorder; or any endocrine disorder with systemic disease which would have impaired overall health and well being (controlled hypo/hyperthyroidism and diabetes mellitus Type II was allowed)
* History or presence of severe psychiatric illness and/or any addictions to drugs, medication or alcohol in the past 3 years
* Diseases for which exogenous hormonal steroids were contraindicated.
* History or presence of any malignancy, except successfully treated non-melanoma skin cancers
* History or presence of cardiovascular or cerebrovascular conditions, thrombosis or thromboembolic disorders
* History or presence of liver, gallbladder or renal disease, epilepsy or classical migraine headaches
* Uncontrolled hypertension
* Women with abnormal cervical smear results
* History or presence of breast cancer, suspicious breast lump or mammographic abnormality
* Known hypersensitivity to any of the ingredients of the trial medication.
* Non-compliance with the screening diary
* Current use of raloxifene, clonidine, veralipride, phytoestrogen extracts
* Drugs known to interfere with the pharmacokinetics of the steroids
* Use of investigational drugs within the past 60 days
* Any disease or condition that was clinically relevant and which, in the opinion of the investigator, would have jeopardized the subject's well being during the course of the trial

Ages: 48 Years to 68 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2004-03-23 (Actual); Primary Completion 2005-11-15 (Actual); Study Completion 2005-11-15 (Actual)

PRIMARY OUTCOMES:
Compare the effect of tibolone (2.5 mg) to transdermal E2/NETA (50/140 mcg) on the vaginal bleeding and spotting rate in healthy postmenopausal women with sexual dysfunction. | Week 13-24 of the in treatment period
Compare the effect of tibolone to E2/NETA on sexual functioning in healthy postmenopausal women with sexual dysfunction. | Week 8-12 and Week 20-24 of the in-treatment period.

SECONDARY OUTCOMES:
Compare the effects of tibolone to E2/NETA on the frequency of satisfactory sexual events, the frequency of sexual fantasies and subjective arousal, scores on the FSFI, FSDS, WHQ and endocrine parameters | Week 8-12 and Week 20-24 of the in-treatment period

REFERENCES:
- [Result] Nijland EA, Weijmar Schultz WC, Nathorst-Boos J, Helmond FA, Van Lunsen RH, Palacios S, Norman RJ, Mulder RJ, Davis SR; LISA study investigators. Tibolone and transdermal E2/NETA for the treatment of female sexual dysfunction in naturally menopausal women: results of a randomized active-controlled trial. J Sex Med. 2008 Mar;5(3):646-56. doi: 10.1111/j.1743-6109.2007.00726.x. PMID 18304284